CLINICAL TRIAL: NCT03908424
Title: Chronic Headache and Chronic Backache Following Unintentional Dural Puncture at Delivery Room
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Alexander Ioscovich, Chair of the Department of Obstetric and Ambulatory Anesthesia, Shaare Zedek Medical Center
Other Study IDs: 0335-18-SZMC
Record Dates: First submitted 2019-04-04; First posted 2019-04-09 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Parturient Who Underwent Epidural Anesthesia During Which an Unintentional Dural Punctur Occurred; Parturient Who Develop a Postdural Puncture Headache; Parturient Who Gave Informed Consent to Participation in the Study
Keywords: PDPH - Post Dural Puncture Headache; chronic headache; chronic backache
MeSH Terms: conditions — Post-Dural Puncture Headache; Headache Disorders | interventions — Blood Patch, Epidural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CONTROL: Parturients who gave birth to a normal birth and did not receive epidural anesthesia.
- Normal Epidural: Parturients who gave birth to a normal birth with epidural anesthesia without an unintentional dural puncture.
- PDPH conservative treatment: Parturients who gave birth to a normal birth with epidural anesthesia and had an unintentional dural puncture, these women were treated conservatively.
- PDPH treated with Blood Patch: . Parturients who had a normal birth with epidural anesthesia and had an unintentional dural puncture and were treated with a blood patch following PDPH.
  Interventions: Other: Epidural Blood patch.

INTERVENTIONS:
Other: Epidural Blood patch. — An epidural blood patch is a surgical procedure that uses autologous blood in order to close one or many holes in the dura mater of the spinal cord, usually as a result of a previous lumbar puncture. A small amount of the patient's blood is injected into the epidural space near the site of the original puncture; the resulting blood clot then "patches" the meningeal leak. An epidural needle is inserted into the epidural space at the site of the cerebrospinal fluid leak and blood is injected. The clotting factors of the blood close the hole in the dura.
  Groups: PDPH treated with Blood Patch

SUMMARY:
he study is a telephone questionnaire. The study will include 400 women, 100 in each group.

OBJECTIVE: To investigate the prevalence of chronic and chronic back pain following PDPH accidental dural puncture during epidyral analgesia for delivery.

1. Parturients who gave birth to a normal birth and did not receive epidural anesthesia.
2. Parturients who gave birth to a normal birth with epidural anesthesia without an unintentional dural puncture.
3. Parturients who gave birth to a normal birth with epidural anesthesia and had an unintentional dural puncture, these women were treated conservatively.
4. Parturients who had a normal birth with epidural anesthesia and had an unintentional dural puncture and were treated with a blood patch following PDPH.

DETAILED DESCRIPTION:
Epidural anesthesia for pain relief during childbirth is performed in about 70% of the parturients in Shaare Zedek Medical Center. The most common complication of epidural analgesia is an unintentional dural puncture occurring in 0.4% -6% of births. Puncture causes acute headache in 70% -80% of cases. The standard treatment is the first stage of conservative treatment of painkillers and caffeine and in the absence of improvement of perform epidural blood patch 24-48 hours after the dural puncture was performed.

There is no widespread support for the literature that a dural puncture with a large diameter needle is a risk factor for the development of chronic headache. For this purpose, we are interested in conducting a study to examine the prevalence of chronic headache and back pain in parturients who underwent epidural anesthesia with a dural puncture to confront parturients who underwent epidural anesthesia without puncturing the dura membrane.

We know that in the years 2017-208 there were about 100 women in the hospital who had a blood patch and a similar number of women who had PDPH and were treated conservatively. From the medical records, we will randomize another 200 mothers, of which 100 were born naturally without epidural anesthesia and another 100 who gave birth to a normal birth with epidural anesthesia without dural puncture.

The study will be conducted using a telephone questionnaire. The telephone questionnaire will be taken at least six months after the epidural anesthesia check if the symptoms are chronic in nature.

Telephone questionnaire carried out four groups of mothers:

1. Parturients who gave birth to a normal birth and did not receive epidural anesthesia.
2. Parturients who gave birth to a normal birth with epidural anesthesia without an unintentional dural puncture.
3. Parturients who gave birth to a normal birth with epidural anesthesia and had an unintentional dural puncture, these women were treated conservatively.
4. Parturients who had a normal birth with epidural anesthesia and had an unintentional dural puncture and were treated with a blood patch following PDPH.

The questionnaire will be performed after receiving informed consent from the patient. Each group will have 100 women.

The questionnaire (attached as an appendix) will examine the prevalence of chronic headache and chronic back pain in these women. Our hypothesis is that in women with PDPH the incidence of chronic headache will be higher.

The statistical comparison between the groups will examine demographic characteristics and characteristics related to frequency of pain, intensity, restriction of daily activity and ways to relieve pain.

Comparisons between the groups for continuous variables will be done with the student t-test and data are presented as mean (standard deviation (SD)), for nonparametric tests with Mann-Whitney test and data are presented as median (interquartile range) ) [range] and for categorical values with Chi-square test and data are presented as number (percentage). A p-values <0.01 will be considered significant due to multiple comparisons. A multivariable regression analysis will be performed to evaluate factors (PDPH, epidural blood patch (EBP), chronic headache, chronic backache) associated with PPD.

ELIGIBILITY:
Inclusion Criteria:

* Parturient who underwent epidural anesthesia during which an unintentional dural punctur occurred.
* Parturient who develop a postdural puncture headache.
* Parturient who gave informed consent to participation in the study.

Exclusion Criteria:

* Parturient without a clear dural hole during operation.
* Parturient who have chronic headaches or migraines.
* Parturient who have chronic back pain.
* Parturient who did not give informed consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who gave birth at Shaare Zedek Medical Center are a tertiary hospital with more than 16,000 births a year. Fifty-five percent of women give birth with epidural anesthesia.
Sampling Method: Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Chronic Headache | At least six months after birth.
  Chronic headache development after PDPH, comparison between different groups. The diagnosis of chronic headache will be done using a questionnaire (attached as an appendix) including the Chronic Pain Grade Questionnaire (Smith et al). The main questions in the questionnaire are the incidence of headache, the severity of the headache, the duration of the problem. Disability Index is also determined by the questions about limiting pain in daily activities.
chronic Backache | At least six months after birth.
  Chronic backache development after PDPH, comparison between different groups. The diagnosis of chronic back pain will be done using a questionnaire (attached as an appendix) including the Low Back Pain Rating Scale (Manniche et al.). The main questions in the questionnaire are the incidence of back pain, severity of back pain, duration of the problem. Disability Index is also determined by the questions about limiting pain in daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Meedical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Loubert C, Hinova A, Fernando R. Update on modern neuraxial analgesia in labour: a review of the literature of the last 5 years. Anaesthesia. 2011 Mar;66(3):191-212. doi: 10.1111/j.1365-2044.2010.06616.x. PMID 21320088
- [Result] Paech M, Banks S, Gurrin L. An audit of accidental dural puncture during epidural insertion of a Tuohy needle in obstetric patients. Int J Obstet Anesth. 2001 Jul;10(3):162-7. doi: 10.1054/ijoa.2000.0825. PMID 15321604
- [Result] Berger CW, Crosby ET, Grodecki W. North American survey of the management of dural puncture occurring during labour epidural analgesia. Can J Anaesth. 1998 Feb;45(2):110-4. doi: 10.1007/BF03013247. PMID 9512843
- [Result] MacArthur C, Lewis M, Knox EG. Accidental dural puncture in obstetric patients and long term symptoms. BMJ. 1993 Apr 3;306(6882):883-5. doi: 10.1136/bmj.306.6882.883. PMID 8490410
- [Result] Smith BH, Penny KI, Purves AM, Munro C, Wilson B, Grimshaw J, Chambers WA, Smith WC. The Chronic Pain Grade questionnaire: validation and reliability in postal research. Pain. 1997 Jun;71(2):141-7. doi: 10.1016/s0304-3959(97)03347-2. PMID 9211475

DOCUMENTS (1):
  • Informed Consent Form (2019-04-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT03908424/ICF_000.pdf